CLINICAL TRIAL: NCT07136246
Title: Research on the Construction of a Prognostic Model for COPD Complicated With Sarcopenic Obesity Based on Bioelectrical Impedance Phase Angle Technology
Brief Title: A Prognostic Model for COPD Complicated With Sarcopenic Obesity Based on Bioelectrical Impedance Phase Angle Technology
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Hospital director, Fudan University
Other Study IDs: COSAT
Record Dates: First submitted 2025-06-29; First posted 2025-08-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenic Obesity; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD with sarcopenic obesity: COPD with sarcopenic obesity based on Bioelectrical Impedance Phase Angle Technology by the enrollment
  Interventions: Device: InBody S10
- COPD without sarcopenic obesity: COPD without sarcopenic obesity based on Bioelectrical Impedance Phase Angle Technology by the enrollment
  Interventions: Device: InBody S10

INTERVENTIONS:
Device: InBody S10 — Bioelectrical Impedance Phase Angle Technology Measured via InBody S10 at six frequencies (1kHz-1000kHz) during each follow-up

SUMMARY:
This study aims to explore the diagnosis, impact, and prognostic factors of COPD complicated with sarcopenic obesity using multi-segment bioelectrical impedance phase angle technology. It seeks to clarify the diagnostic value and efficacy of body composition analysis in specific populations, analyze the relationship between phase angle and COPD severity as well as quality of life, investigate its predictive role for adverse outcomes, and reveal the effects of inflammation and metabolic disorders in sarcopenic obesity. The goal is to provide a basis for early screening and precise intervention to improve patient prognosis.

DETAILED DESCRIPTION:
The primary objective of this study is to use multi-segment bioelectrical impedance phase angle technology to explore the diagnosis, impact, and prognostic factors of COPD complicated with sarcopenic obesity. The study aims to clarify the diagnostic value and efficacy of body composition analysis in specific populations, analyze the relationship between phase angle and COPD severity as well as quality of life, investigate its predictive role for adverse outcomes, and reveal the effects of inflammation and metabolic disorders in sarcopenic obesity. The goal is to provide a basis for early screening and precise intervention to improve patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 65 years;
2. Ability to complete physical activity assessments and pulmonary function tests;
3. Complete medical records, willingness to adhere to follow-up arrangements, and provision of adverse event reports via telephone or outpatient visits, with signed informed consent;
4. COPD diagnosis based on the American Thoracic Society (ATS)/European Respiratory Society (ERS) GOLD definition, with a post-bronchodilator FEV1/FVC ratio < 0.70, current or former smokers with a smoking history of ≥10 pack-years.

Exclusion Criteria:

1. Severe cognitive impairment or hand deformities (e.g., rheumatoid arthritis) preventing body composition measurements;
2. Incomplete clinical or follow-up data or unwillingness/inability to undergo regular follow-up;
3. Severe systemic edema;
4. Presence of cardiac pacemakers or significant metal implants that may interfere with measurements;
5. Voluntary withdrawal for any reason, including loss to follow-up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The elderly COPD patients measured with bioelectrical impedance phase angle technology
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
Changes in pulmonary function | 6, 12, and 24 months
  FEV1%
COPD Assessment Test (CAT) | 6, 12, and 24 months
  The COPD Assessment Test (CAT) is a short, validated questionnaire used to measure the impact of COPD symptoms on a patient's daily life and health status. It consists of 8 simple questions, each scored from 0 to 5, with a total range of 0-40.Higher CAT scores = Worse COPD symptoms & greater disease burden
Body composition | 6, 12, and 24 months
  Segmental phase angles measured via bioelectrical impedance analysis
Dyspnea Scale | 6, 12, and 24 months
  The Modified Medical Research Council(mMRC) scale is a simple questionnaire used to assess the severity of breathlessness, primarily in respiratory diseases like COPD.range from 0-4 .Grading Criteria:Grade 1: Short of breath when walking fast or climbing a slight hill.Grade 2: Walk slower than peers or need to stop occasionally due to breathlessness.Grade 3: Stop to breathe after walking ~100 meters or a few minutes on level ground.Grade 4: Too breathless to leave home, or breathless while dressing/undressing.A higher mMRC grade correlates with greater dyspnea severity and more pronounced symptoms."

SECONDARY OUTCOMES:
Acute exacerbations | 6, 12, and 24 months
  An acute exacerbation of chronic obstructive pulmonary disease (AECOPD) is defined as:An acute worsening of respiratory symptoms that results in additional therapy.
Hospitalizations | 6, 12, and 24 months
  Frequency of hospitalizations
Mortality | 24 months
  Mortality based on Mal-Nutritional Status
CBC | 6, 12, and 24 months
  Serum level of WBC (ELISA)
CRP | 6, 12, and 24 months
  Serum level of C-Reactive Protein (ELISA)
albumin | 6, 12, and 24 months
  Serum level of albumin
IL-6 | 6, 12, and 24 months
  Serum level of Interleukin-6
TNF-α | 6, 12, and 24 months
  Serum level of Tumor Necrosis Factor-alpha

CONTACTS AND LOCATIONS:
Overall Officials: Yinggang Zhu, MD, PhD, Principal Investigator — Huadong Hospital
Locations (1):
- Huadong hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT07136246/Prot_SAP_001.pdf